CLINICAL TRIAL: NCT03540173
Title: A New Intubation Discomfort Score Identified Patients' Painfulness During Unsesated Colonoscopy
Brief Title: Discomfort Score Identifies Painfulness During Unsedated Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: KY20180128-1
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Risk Factors Associated With Painful Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: In the training cohort, we evaluated the impact of patient-related factors on the pain during the colonoscopy. In univariatelogistic regression analysis, All factors associated with the pain during colonoscopy (p<0.1) were included in multivariate analysis.
- Validation group: The validation cohort was used to verify the intubation discomfort score.

SUMMARY:
Some patients felt no pain or only mild discomfort with the unsedated colonoscopy. However, unsedated colonoscopy was thought to be an option for some but not for all. If we could able to identify which patients at high risk for painful colonoscopy in preoperational stage, targeted administration of sedatives or special techniques to these patients would be an attractive option.

DETAILED DESCRIPTION:
Here we prospectively collected the data during colonoscopy and investigated the possible risk factors associated with painful colonoscopy by using a step-wise multivariate regression model. Furthermore we developed a novel point score to predict whether the patients at high risk for painful colonoscopy and targeted offer an appropriate method of colonoscopy or with the aid of special techniques to help the completion of procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent unsedated colonoscopy

Exclusion Criteria:

* (1) no bowel preparation or colon cleansing by enema only; (2) no need to reach cecum; (3) prior finding of severe colon stenosis or obstructing tumor; (4) history of colectomy; (5) unstable hemodynamics; (6) pregnant; (7) unable to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were prescribed polyethylene glycol electrolyte for bowel preparation according to the preference of physicians. They were asked to drink the first 2L of PEG4000e at19:00-20:00 PM on the night before colonoscopy within 2 hours. Then, on the day of the examination, patients were asked to take the remaining 2L 5 hours before the procedure. Patients were encouraged to drink more clear liquids after purgatives for adequate hydration before colonoscopy. In addition, patients were instructed to have a regular meal for lunch and only liquid diets for dinner the day before the operation.
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
The anxiety status | 1 year
  Hospital Anxiety and Depression Scale (HAD)

SECONDARY OUTCOMES:
Abdominal pain | 1 year
  Abdominal pain evaluated by a previously validated 4-point verbal rating scale (no, slight, moderate, severe pain)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi